CLINICAL TRIAL: NCT06353477
Title: Use of EPs®7630 in Hand, Foot and Mouth Disease
Brief Title: Hand, Foot, and Mouth Disease: Could EPs®7630 be a Treatment Option
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Principal Investigator, Murat Sutcu, Prof Dr, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EOU 2019-10
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Hand, Foot, and Mouth Disease
Keywords: Hand, foot, and mouth disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Intervention Model Description: EPs® 7630 is an extract from the roots of Pelargonium sidoides, drug-extract ratio 1 : 8-10, extraction solvent ethanol 11% (w/w). The patients were divided into two groups: (i) group 1 received herbal drug EPs® 7630 by oral route [Umca® solution; (3x10 drops; between 1-5 years of age, 3x20 drops; 6-12 years of age, 3x30 drops for children >12 years of age)] for 7 days and (ii) group 2 (control group) did not receive any herbal medication. The medication was administered orally, at least 30 minutes before or after meals. Patients in both groups were prescribed paracetamol (10 mg/kg/dose, 4 times a day, maximum 4,000 mg/day.) as an antipyretic agent. Temperature measurement was made at home and in the hospital via the axillary route.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPs® 7630 group (Active Comparator): The patients were divided into two groups: (i) group 1 received herbal drug EPs® 7630 by oral route [Umca® solution; (3x10 drops; between 1-5 years of age, 3x20 drops; 6-12 years of age, 3x30 drops for children >12 years of age)] for 7 days.
  Interventions: Drug: EPs® 7630
- control grup (No Intervention): Control group did not receive any herbal medication.

INTERVENTIONS:
Drug: EPs® 7630 — EPs® 7630 is an extract from the roots of Pelargonium sidoides, drug-extract ratio 1 : 8-10, extraction solvent ethanol 11% (w/w). The patients were divided into two groups: (i) group 1 received herbal drug EPs® 7630 by oral route [Umca® solution; (3x10 drops; between 1-5 years of age, 3x20 drops; 6-12 years of age, 3x30 drops for children >12 years of age)] for 7 days and (ii) group 2 (control group) did not receive any herbal medication. The medication was administered orally, at least 30 minutes before or after meals. Patients in both groups were prescribed paracetamol (10 mg/kg/dose, 4 times a day, maximum 4,000 mg/day.) as an antipyretic agent. Temperature measurement was made at home and in the hospital via the axillary route.
  Other Names: Group 1
  Arms: EPs® 7630 group

SUMMARY:
This randomized controlled study aims to evaluate the effectiveness and safety of the pharmaceutical extract EPs® 7630 from P.sidoides in treating hand, foot, and mouth disease in children. The study will investigate the impact of EPs® 7630 on the severity of the disease over a specific period and its effects on hospitalization rates and potential complications. This research aims to contribute to the treatment of hand, foot, and mouth disease in children.

DETAILED DESCRIPTION:
Study design This multicenter randomized controlled study was conducted between June 2019- June 2022 in 8 centers in Turkey. These centers were hospitals of reference that provided tertiary care services. The clinical study protocol was approved by the Eskisehir Osmangazi University. This clinical study protocol was approved by the Eskisehir Osmangazi University Interventional Research Ethics Committee with the number 2019-10 and conducted in accordance with the World Medical Association's Declaration of Helsinki and on Good Clinical Practice compliance. This study was conducted with the approval of the Turkish Medicines and Medical Devices Agency Written informed consent was obtained from parents of all patients included in the study.

Study participants and clinical management All of pediatric patients who were examined by a pediatrician and diagnosed with HFMD and start of the symptoms in last 48 hours (either fever or enanthems or exanthem) were offered trial participation. Patients whose complaints lasted more than 48 hours, those whose families stated that they were unable to comply with follow-ups, those did not give informed consent, those taking another antiviral or supportive treatment, those who had used antibiotics in the previous 1 month, those with a history of immunodeficiency or a family history of immunodeficiency, and those with a previous history of anaphylaxis with any supplement or drug, any chronic disease, or skin lesion were not included in the study.

At the first admission, the duration of the patients' complaints, the distribution of the lesions in the body, and the fever status were recorded. Parents were asked to rate the severity of the child's restlessness, inappetence, and sleeplessness status on a scale of 0-10.

Participants were assigned 1:1 to one of two trial arms by a local research team member using a centralized computerized randomization system (RAND2 software, The MathWorks Inc, Natick, United States, contractually managed by the data management team). Lists in four blocks were added to the automatic online randomization system to ensure a homogeneous distribution of the groups in both study centers. On the basis of the power calculations of similar studies, a minimum sample size of 80 per group was calculated to give a 90% probability (power) of producing a significant finding. Overall, 120 patients were designated for the for each group that considering that there may be losses in the study.

All patients were followed up twice more, 48 hours after the first admission and on the 5th-7th days. Another phone evaluation was conducted for those with continued complaints from the previous visit. During these visits, the patient's fever status, restlessness, inappetence, and sleeplessness scores were asked again of their parents and recorded. Patient medication adherence and drug side effects were evaluated. After the patient's recovery, the total duration of the disease and the duration of restlessness, inappetence, and sleeplessness were recorded. Patients who were hospitalized or developed complications were noted.

Intervention EPs® 7630 is an extract from the roots of Pelargonium sidoides, drug-extract ratio 1 : 8-10, extraction solvent ethanol 11% (w/w). The patients were divided into two groups: (i) group 1 received herbal drug EPs® 7630 by oral route [Umca® solution; (3x10 drops; between 1-5 years of age, 3x20 drops; 6-12 years of age, 3x30 drops for children >12 years of age)] for 7 days and (ii) group 2 (control group) did not receive any herbal medication. The medication was administered orally, at least 30 minutes before or after meals. Patients in both groups were prescribed paracetamol (10 mg/kg/dose, 4 times a day, maximum 4,000 mg/day.) as an antipyretic agent. Temperature measurement was made at home and in the hospital via the axillary route.

ELIGIBILITY:
Inclusion Criteria:

-Patients diagnosed with Hand, foot, and mouth disease

Exclusion Criteria:

* Patients whose complaints lasted more than 48 hours
* Unable to comply with follow-ups,
* Did not give informed consent,
* Another antiviral or supportive treatment,
* Use antibiotics in the previous 1 month,
* A history of immunodeficiency or a family history of immunodeficiency,
* A previous history of anaphylaxis with any supplement or drug,
* Any chronic disease, or skin lesion -

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
the patient's fever status, restlessness, inappetence, and sleeplessness scores | All patients were followed up twice more, 48 hours after the first admission and on the 5th-7th days.
  score

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Medicine Faculty Hospital, Esenyurt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
EOU 2019-10
Supporting Information: Study Protocol
Time Frame: March 2024- June 2024
Access Criteria: researchers
URL: https://www.cocukenfeksiyondernegi.org/

REFERENCES:
- [Background] Miller GD, Tindall JP. Hand-foot-and-mouth disease. JAMA. 1968 Mar 4;203(10):827-30. No abstract available. PMID 5694203
- [Derived] Sutcu M, Kara M, Yildiz F, Kilic O, Tural Kara T, Akkoc G, Buyukcam A, Elmas Bozdemir S, Ozgur Gundeslioglu O, Gul D, Iseri Nepesov M, Kara A. Hand, foot, and mouth disease: could EPs(R) 7630 be a treatment option? A prospective randomized open-label multicenter clinical study. Front Pediatr. 2024 May 20;12:1274010. doi: 10.3389/fped.2024.1274010. eCollection 2024. PMID 38832001
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/5694203/